CLINICAL TRIAL: NCT07166913
Title: Enhancing Stakeholder Engagement in Pediatric Research
Brief Title: Enhancing Engagement of Partners in Research
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 24-01851; SOE-2022C2-28894 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2025-09-09; First posted 2025-09-11 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stakeholder Engagement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Strategies (Experimental): Subjects assigned to the Enhanced Strategies arm will receive a toolkit of enhanced stakeholder engagement strategies.
  Interventions: Behavioral: Toolkit
- Standard Practice (No Intervention): No Intervention. Participants will continue to implement standard practices used by investigator

INTERVENTIONS:
Behavioral: Toolkit — The toolkit contains information regarding enhanced stakeholder engagement strategies. The toolkit includes guidance materials, checklists, and templates/ sample materials, to increase stakeholder engagement in the research. This includes guidance on setting up a stakeholder advisory board (SAB) and ensuring literacy- and language- sensitivity of participant-/stakeholder-facing materials.
  Arms: Enhanced Strategies

SUMMARY:
The purpose of this study is to examine the implementation and effectiveness of a bundle of engagement strategies for pediatric patient centered outcomes research (PCOR) studies. The study aims to examine the effectiveness of a "bundle" of enhanced engagement strategies on improved stakeholder engagement and study protocol indicators (including improved language access, meeting recruitment/retention goals) compared to standard practice.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, PIs must oversee a study that meets the following criteria:

1. Studies who either have not started enrollment or are within 1-3 months of the start of enrollment, and within the 25% ceiling for % recruitment target.
2. Studies that have started enrollment must be no further than 25% of projected enrollment timeline of the study (with at least 6 months remaining for enrollment).
3. Target n>50 participants in study.
4. At least 10 stakeholder partners part of study. The PI's must also be ≥18 years old;

In order for study stakeholders to be eligible to participate in this study, an individual must meet all of the following criteria:

1. >=12 years old;
2. Ability to speak either English, Spanish, or Chinese, and;
3. Part of the study team or serving in an advisory capacity to the study team

The same criteria as that used for stakeholder and PI eligibility applies to Key informant (KI) interviews.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Not able to complete 6 month follow-up assessment
2. Children who are wards/foster children
3. Not able or willing to provide consent.
4. Concurrent enrollment in another study that is part of this research project.

In addition, PI's who meet the following criteria will be excluded from participation in this study:

1. A lot of experience with stakeholder engagement (based on screener survey question)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Research Engagement Survey Tool (REST) stakeholder engagement score | Month 6
  This tool consists of 32 items and assesses engagement across 8 domains, using a 5-point Likert scale for each item. The 8 domains include: 1) focus on community perspectives and determinants of health, 2) partner input, 3) partnership sustainability, 4) fostering co-learning, capacity building and co-benefit, 5) building on strengths and resources, 6) facilitating collaborative, equitable partnerships, 7) involving partners in the dissemination process, and 8) building and maintaining trust. Engagement principle (EP) scores are calculated as an average of non-missing items. The 8 means are used to calculate the overall stakeholder engagement score. Higher scores indicate higher degree of stakeholder engagement.

SECONDARY OUTCOMES:
Patient Engagement in Research Scale (PEIRS) stakeholder engagement score | Month 6
  The scale consists of 22 items and assesses engagement across seven domains, using a 5-point Likert scale for each item. The 7 domains include: 1) procedural requirements, 2) convenience, 3) contributions, 4) team environment and interaction, 5) support, 6) feel valued, and 7) benefits. The total score is calculated by summing the scores for each item and dividing by the maximum possible score. This result is then multiplied by 100 to get a score out of 100. Higher scores indicate a greater degree of meaningful patient engagement.
Reading grade level of written materials | Month 6
  Mean of 5 readability formulas (Flesch Reading Ease, Flesch-Kincaid, Simple Measure of Gobbledygook (SMOG), Gunning Fog, Forcast). Lower score reflects lower reading grade level.
Patient Education Materials Assessment Tool (PEMAT) score | Month 6
  Consists of Understandability (19 items) and Actionability (7 items) subscales. Scoring is as follows: (Total points / possible points yields) x100 = Score %. Higher score reflects greater understandability / actionability.

CONTACTS AND LOCATIONS:
Overall Officials: H. Shonna Yin, MD, MS, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Hsiang.Yin@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Hsiang.Yin@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.